CLINICAL TRIAL: NCT01356108
Title: Implantation of the SAPIEN™ Transcatheter Heart Valve (THV) in the Pulmonic Position
Brief Title: Pulmonic Valve REplacement Multi-discIpline EMEA Registry
Acronym: PREMIER
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010-11
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Regurgitation; Pulmonary Insufficiency; Pulmonary Stenosis
Keywords: Conduit; Pulmonic; Stenosis; Regurgitation; Dysfunctional
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Respiratory Insufficiency; Pulmonary Valve Stenosis; Constriction, Pathologic; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Transcatheter Pulmonic Valve Replacement (TPVR) (Edwards SAPIEN™ THV) — The Edwards SAPIEN™ THV is a biological heart valve manufactured with treated bovine pericardial tissue that is mounted into a balloon expandable stainless steel open cell stent. The Edwards SAPIEN™ THV is available in two sizes (23 and 26mm) and is designed for transcatheter implantation in patients with regurgitant pulmonary valved conduit with or without stenosis. This device is commercially available and is used according the current IFU.

SUMMARY:
The purpose of this registry is to retrospectively and prospectively obtain clinical data in consecutively treated patients, in order to demonstrate that the commercially available Edwards SAPIEN Valve with the RF3 delivery system is a safe and effective treatment for patients with pulmonary regurgitation or stenosis.

DETAILED DESCRIPTION:
Consecutive patient data should be collected at discharge, 6 months, 12 months and 2-5 years post-implant.

ELIGIBILITY:
Inclusion Criteria:

- Symptomatic with a regurgitant or stenotic pulmonary valved conduit.

Exclusion Criteria:

* Angiographic evidence of coronary artery compression.
* RV-PA pulmonary conduit size that is either too large or too small to accommodate the SAPIEN THV.
* Thrombus or intracardiac mass in the right atrium, right ventricle, and/or pulmonic valve.
* Severe coagulation problems and/or unable to tolerate anticoagulation/antiplatelet therapy.
* Active bacterial endocarditis or other active infections.
* Illeofemoral venous stenosis that may prevent the placement of the introducer sheath and/or central venous vascular tortuosities that may prevent advancement of the delivery system to the heart or into the pulmonary artery.
* Presence of any prosthetic valve in the tricuspid position.
* Unstable coronary artery disease-related angina.
* Placement of the SAPIEN THV in pregnant females.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All symptomatic patients with a regurgitant or stenotic pulmonary valved conduit treated by implantation of the Edwards SAPIEN™ THV.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months
  Procedure/Device Success and Freedom from device or procedure related death

SECONDARY OUTCOMES:
Safety and Effectiveness | 6 Months
  Freedom from device or procedure related SAE and functional improvement

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ewert, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (16):
- University Hospital Leuven, Leuven, Belgium
- Germany (4):
  - Herz und Diabeteszentrum NRW, Bad Oeynhausen
  - German Heart Institute Berlin, Berlin
  - Deutsches Herzzentrum München, München
  - Universitätsklinikum Münster, Münster
- Mater Misericordiae University Hospital, Dublin, Ireland
- Schneider Children's Medical Center of Israel, Petach Tikvah, Israel
- Italy (2):
  - Ospedale Bambino Gesù, Rome
  - Policlinico San Donato, San Donato Milanese
- The Cardinal Stefan Wyszyński Institute of Cardiology, Warsaw, Poland
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Centre, Riyadh
  - Prince Sultan Cardiac Centre, Riyadh
- Mehmet Akif Ersoy Thoracic & Cardiovascular Surgery, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - Royal Brompton Hospital, London
  - The Heart Hospital, London
  - Manchester Royal Infirmary, Manchester